CLINICAL TRIAL: NCT06200675
Title: How Best to Understand and Intervene With State Shame and Self-criticism: A Randomised Clinical Trial Comparing Two Theoretical Perspectives
Brief Title: Understanding and Intervening With State Shame and Self-criticism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, Allison Kelly, Associate Professor, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 45443
Record Dates: First submitted 2023-12-19; First posted 2024-01-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Self-Criticism
Keywords: Self-compassion; Compassion; Online single-session intervention

STUDY DESIGN:
Intervention Model Description: 1/3 of the study participants (anticipated n=116) will be randomly assigned to the self-compassion intervention group, 1/3 of the participants (anticipated n=116) will be placed into the logic-based intervention group, and 1/3 of the study participants (anticipated n=116) will be placed into the control group.
Who Masked: Participant
Masking Description: The participant will not know prior to their study participation that there are three different study conditions, and they will not find out which condition they were randomized to until the end of their study participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compassion-based intervention (Experimental): Participants assigned to this intervention will be asked to engage in one brief (10-15 minute) online compassion-focused exercise, where they will be asked to connect to their inner compassionate self. They will be asked to stay connected to that feeling while rereading what they wrote about their feelings of shame and imagining it was someone else who wrote it. Participants will then be asked to write a compassionate response to themselves. Participants will then be asked to reread this response while remaining connected to their compassionate self.
  Interventions: Other: Compassion-based intervention
- Logic-based intervention (Experimental): Participants assigned to this intervention will be asked to engage in one brief (10-15 minute) online logic-based exercise that was adapted from a thought record (Greenberger & Padesky, 1995), which is often completed during cognitive behavioural therapy (CBT) treatment. Participants will be asked to reread what they wrote about their feelings of shame and chose a thought central to their shame to use for this exercise. Participants will be asked to generate evidence for and against their chosen thought, and then generate a more balanced thought. After the exercise, participants will be asked to reread their newly generated more balanced thought.
  Interventions: Other: Logic-based intervention
- Placebo control condition (Active Comparator): Participants assigned to this condition will be asked to listen to a portion of an audio recording of "The Hobbit" (Tolkien, 2009) and then re-read what they wrote about their feelings of shame. They will then be asked to write a reflection about the thoughts and feelings arising from doing so. They will then be asked to re-read what they wrote in this reflection.
  Interventions: Other: Placebo control condition

INTERVENTIONS:
Other: Compassion-based intervention — Participants assigned to this intervention will be asked to engage in one brief compassion-focused exercise, where they will be asked to be asked to connect to their inner compassionate self. They will be asked to stay connected to that feeling while rereading what they wrote about their feelings of shame and imagining it was someone else who wrote it. Participants will then be asked to write a compassionate response to themselves. Participants will then be asked to reread this response while remaining connected to their compassionate self.
  Arms: Compassion-based intervention
Other: Logic-based intervention — Participants assigned to this intervention will be asked to engage in one brief (10-15 minute) online logic-based exercise that was adapted from a CBT thought record. Participants will be asked to reread what they wrote about their feelings of shame and chose a thought central to their shame to use for this exercise. Participants will be asked to generate evidence for and against their chosen thought, and then generate a more balanced thought. After the exercise, participants will be asked to reread their newly generated more balanced thought.
  Arms: Logic-based intervention
Other: Placebo control condition — Participants assigned to this intervention will be asked to listen to an audio recording of "The Hobbit" and then re-read what they wrote about their feelings of shame. They will then be asked to write a reflection about the thoughts and feelings arising from doing so. They will then be asked to re-read what they wrote in this reflection.
  Arms: Placebo control condition

SUMMARY:
The goal of this clinical trial is to compare the momentary effects of a one-session intervention (compassion-based, logic-based, or placebo control) on individuals with high or low trait self-criticism. The main questions it aims to answer are:

After a momentary shame induction, will a compassion-based intervention and a logic-based intervention both be more beneficial than a placebo control condition in terms of therapeutic outcomes?

Will the compassion-based intervention most effectively increase soothing affect, state self-compassion, and state self-reassurance?

Will the effects of these two interventions (1) differ as a function of the individual's trait self-criticism, and (2) will this be due to differing indirect effects of the intervention on safe/soothed feelings based on trait self-criticism?

Participants will first complete a set of baseline measures. Two to seven days later, they will be randomly assigned to one of three study conditions (i.e., compassion-based, logic-based, placebo control) after a brief shame induction. Participants will be asked to complete a set of questionnaires both before and after the shame induction as well as post-intervention.

This research will help us understand how best to intervene with the shame and self-criticism.

DETAILED DESCRIPTION:
This clinical trial consists of a two-part online study. Part 1 of this study collects baseline measures and screen out ineligible participants. Part 2 of this study will compare the momentary effects of a brief (10-15 minute) one-session online intervention (compassion-based, logic-based, or placebo control) after a shame induction. Participants assigned to the compassion-based intervention will be asked to engage in a self-compassion exercise, where they will be asked to write about and experience their feelings while connecting to their compassionate self. Participants assigned to the logic-based intervention will be asked to engage in a logic-based exercise that was adapted from a thought record often completed during CBT treatment. Participants assigned to the placebo control condition will be asked to listen to a portion of an audio recording of "The Hobbit." All conditions will involve audio recordings, and all participants will be asked to re-read what they wrote about their shame, engage in a writing task, and then re-read what they wrote during the intervention writing task.

ELIGIBILITY:
Inclusion Criteria for SONA participants:

* Participants will be UWaterloo undergraduate students with a SONA account.
* Participants must be able to listen to audio clips (either via device speakers or with headphones) during their study participation.

Inclusion Criteria for Prolific participants:

* Participants will be adults (i.e., 18-64 years of age) with a Prolific account.
* Participants must be able to listen to audio clips (either via device speakers or with headphones) during their study participation.
* Prolific participants must also be first language English speakers.

Exclusion Criteria:

All exclusions will only be made prior to randomization of experimental conditions in Part 2 to abide by Consort guidelines for randomized controlled trials.

1. Any duplicate survey completions from the same participant for the same study survey, as indicated by their embedded ID code in their Qualtrics data, will be excluded from analysis. For Part 1, the most complete survey completion for each participant will be retained. For Part 2, the most complete survey completion for each participant will also be retained unless the participant has begun the shame induction exercise. If a participant in Part 2 has begun the shame induction and then completes another submission, they will be excluded.
2. Participants who do not complete Part 1 measures required for primary hypotheses will also be excluded from analyses (specifically, participants who do not complete the measures of trait self-criticism and trait self-compassion).
3. Participants who complete Part 1 but are not randomized to a condition in Part 2, will be excluded from analyses related to Part 2 variables. We will run ANOVAs and/or non-parametric Kruskal Wallis tests with continuous baseline data as the DVs to test if there are any significant differences between participants who do Part 2 and those who do not. We will also run Fisher-Freeman-Halton exact tests on categorical baseline data to test if there are any significant differences between participants who do Part 2 and those who do not.
4. Participants who respond to several scales within the same survey with overly consistent responses (i.e., appear to click the same response for every scale item, even though some are reverse scored, assessed via testing of scale variances) may be excluded from analyses involving that survey. Their data from other surveys will still be retained for other analyses.
5. Participants who complete a survey in an unreasonably short or long amount of time compared to the average participant may be excluded from analyses involving that survey. Their data from other surveys will still be retained for other analyses.
6. Participants who fail half or more of the attention checks in Part 1, and the first attention check prior to randomization in Part 2 will be excluded from the data.
7. Participants who were ineligible or withdrew consent will also be excluded from the data.
8. Prolific participants who could not complete the Captcha Verification question or fail one or both of the two bot check questions will also be excluded from the analyses.
9. We will inspect the distribution of scores on trait self-criticism and consider excluding extreme outliers with very low or very high scores.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
State Shame and Guilt Scale (shame subscale) | Immediately pre-shame induction, immediately after the shame induction, immediately after the intervention
  Self-report questionnaire with 5 items on a 5-point Likert scale (scored 1-5). Mean scores range from 1-5, with higher scores indicating greater momentary feelings of shame.
Momentary self-criticism | Immediately pre-shame induction, immediately after the shame induction, immediately after the intervention
  Self-report questionnaire with 5 items on a 5-point Likert scale (scored 1-5). Mean scores range from 1-5, with higher scores indicating greater momentary self-criticism.
Self-Assessment Manikin (Arousal and Pleasure subscales only) | Immediately pre-shame induction, immediately after the shame induction, immediately after the intervention
  Self-report measure with 1 item assessing arousal and 1 item assessing pleasure, on a pictorial 9-point Likert scale (scores ranging from 1-9). Items are scored individually, and higher scores indicate greater degrees of arousal or pleasure.

SECONDARY OUTCOMES:
Soothing affect | Immediately after the intervention
  This adapted measure consists of the Serenity Subscale of the PANAS-X, the Safe/Warmth Positive Affect Subscale of the Types of Positive Affect Scale, and researcher-generated items). Self-report questionnaire consists of 13 items on a 5-point Likert scale (scored 1-5). Mean scores range from 1-5, with higher scores indicating higher degrees of soothing affect.
State self-compassion assessed via Compassionate Engagement and Action Scale (adapted self-compassion subscale) | Immediately after the intervention
  Self-report measure consisting of 13 items on a 10-point Likert scale (scored 1-10), with higher scores indicating greater state self-compassion.
State self-compassion assessed via State Self-Compassion Scale (adapted) | Immediately after the intervention
  Self-report measure consisting of 6 items rated on a 5-point Likert scale (scored from 1-5). Mean scores range from 1-5, with higher scores indicating greater state self-compassion.
Self-reported reassurance (researcher-generated) | Immediately after the intervention
  Self-report measure consisting of 4 items assessed on a 5-point Likert scale (scored 1-5). Mean scores range from 1-5, with higher scores indicating greater self-reassurance.

CONTACTS AND LOCATIONS:
Overall Officials: Allison C. Kelly, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenberger, D., & Padesky, C. A. (1995). Mind over mood: A cognitive therapy treatment manual for clients. Guilford Press.
- [Background] Tolkien, J. R. R. (2009). The Hobbit (E-book ed.). HarperCollins.